CLINICAL TRIAL: NCT05596617
Title: Safety and Efficacy of Drugs Given Off-label for COVID-19
Brief Title: Safety and Efficacy of Medications COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Miguel Sanchez Garcia, Director Critical Care, Hospital San Carlos, Madrid
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Meds Off-label
Record Dates: First submitted 2022-10-20; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Severe Covid-19
Keywords: Covid-19; Adverse events; Organ dysfunction; Mortality
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: quasi-experimental
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of care management of severe Covid-19 patients
- Oral bedtime melatonin (Experimental): Standard of care with oral bedtime melatonin
  Interventions: Drug: Oral bedtime melatonin

INTERVENTIONS:
Drug: Oral bedtime melatonin — Different doses of oral bedtime melatonin
  Other Names: Standard of care
  Arms: Oral bedtime melatonin

SUMMARY:
We performed a quasi-experimental open-label pragmatic study alternating standard of care (SOC) and oral bedtime melatonin (OBM) at different high doses over 4 consecutive time periods enrolling all consecutive RT-PCR SARS-CoV-2 severe Covid-19 admissions.

DETAILED DESCRIPTION:
The 4 successive study time periods spanned from March 2020 to April 2021 and included: 1) standard of care (SOC) (C1), 2) SOC + oral bedtime melatonin (OBM) (T1), 3) SOC (C2), and 4) SOC + OBM (T2). During T1, 3 consecutive subgroups received 50 mg, 100 mg and 200 mg OBM. During T2, 100 mg OBM was given. Melatonin was administered from ICU admission to hospital discharge or death.

The main objectives were occurrence of predefined severe adverse events (SAEs), Sequential Organ Failure Assessment (SOFA) scores and day-30 (D30) and 90 (D90) mortality. Study subjects were followed for modified Rankin scale (mRS) at 30 days after the last OBM dose or hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Positive RT-PCR for SARS-CoV-2

Exclusion Criteria:

* Anticipated death within 48 hours or paliative care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Severe adverse events | From date of inclusion until date of hospital discharge or death
  predefined severe adverse events
Organ dysfunction | On days 1, 4, 7, 14 and 30 since first dose of melatonin
  Sequential organ failure assessment score
Mortality | On days 30 and 90 since first dose of melatonin
  From date of inclusión to date of day 30 and day 90 mortality

SECONDARY OUTCOMES:
Length of stay | Date of inclusion until date of ICU and hospital discharge or death
  Length of ICU and hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Fernandez-Tresguerres, MD.PhD, Study Chair — Universidad Complutense Madrid
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Yes, although after publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication
Access Criteria: Privision of an analysis plan